CLINICAL TRIAL: NCT00107757
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 50mcg and 100mcg for 2 Weeks in Pediatric Subjects Ages 2 to <12 Years With Seasonal Allergic Rhinitis (SAR)
Brief Title: Seasonal Allergic Rhinitis In Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR100010
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: pediatric; Seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal

INTERVENTIONS:
Drug: GW685698X

SUMMARY:
The purpose of this study is to determine if the investigational drug is effective and safe in children with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of seasonal allergic rhinitis.
* Adequate exposure to seasonal (Spring/Summer) allergen prevalent to the geographic area.

Exclusion criteria:

* Have significant concomitant medical conditions.
* Use of corticosteroids, other allergy meds during the study.
* Have abnormal ECG or laboratory abnormality.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 576
Dates: Start 2005-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Improvement in daily, reflective total nasal symptom scores after 2 weeks of treatment in subjects ages 6 to <12 years.

SECONDARY OUTCOMES:
Improvement in AM, pre-dose, instantaneous total nasal symptom scores after 2 weeks of treatment, overall evaluation of response to therapy after 2 weeks of treatment for subjects ages 6 to <12 years.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (61):
- United States (61):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Cudahy, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, North Andover, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Cranberry Township, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR100010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register